CLINICAL TRIAL: NCT02635113
Title: Falls Prevention Using a Gait-Synchronized Vibration System
Brief Title: Falls Prevention: Gait-Synchronized Vibration System
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: NYU Langone Health (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-00617
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Sensory Deficits
Keywords: balance; gait; falls; sensory deficits; vibration; visual acuity; dizziness; postural control; proprioceptive function; stereoacuity; depth perception; vestibular dysfunction
MeSH Terms: conditions — Dizziness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD Shoe (Experimental): 40 subjects will wear the shoe in order to test abnormal gait patterns that increase likelihood of falls and the effectiveness of a gait synchronized vibration system to plantar surface to reduce fall risk.
  Interventions: Device: Gait Synchronized Vibration System

INTERVENTIONS:
Device: Gait Synchronized Vibration System — A wearable vibratory shoe that delivers stimulus to the soles that is synchronized with step resulting in improved gait.The shoe consists of two externally mounted vibration units (tactors). The vibration units allow for variation of both frequency and amplitude of stimulation independently. Using the pressure sensors and timing data, gait velocity, cadence, swing time, stance phase and double support time will be analyzed to assess features of their gait performance during the Dynamic Gait Index with and without vibratory stimuli.
  Other Names: PD shoes

SUMMARY:
The purpose of this study is to develop an abnormal gait detection algorithm and a vibratory stimulation system on a lower limb to improve gait stability and prevent falls. The investigators want to detect, assess and communicate fall risk indicators obtained via the shoe sensors, and assess effectiveness of a gait synchronized vibration system to the plantar surface in reducing fall risk.The system consists of a gait measurement module, an abnormal gait detection module, and a vibratory stimulation module.

DETAILED DESCRIPTION:
Forty (40) Individuals with decreased confidence in ambulatory scores (<80%) as per the Activities Specific Balance Confidence questionnaire, will undergo functional assessments for visual (Snellen chart, Humphrey Visual Field Testing, Gaze Stabilization test, depth perception evaluation), vestibular (Dizziness Handicap Inventory, Head Thrust test) and proprioceptive (Balance Master, Berg Balance Scale, Joint Position Sense) impairments, to evaluate factors which might contribute to increased falls risk.

Participants will be asked to walk return for a second visit and to walk with a shoe sensor and gait synchronized vibratory stimulus under conditions of (1) Baseline performance on the Six Minute Walk test (2) Performance on the Six Minute Walk test and Dynamic Gait Index without vibratory stimulus (3) Performance on the Six Minute Walk test and Dynamic Gait Index with vibratory stimulus.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 65 or greater.
2. Low balance confidence (scores <80%) on the ABC Balance Confidence Scale
3. Berg Balance Scale (BBS) scores between 21 (moderate fall risk) and 56 (low fall risk).

Exclusion Criteria:

1. No internal implantable device (i.e. Pacemaker, Intrathecal Baclofen Pump)
2. Significant painful arthritis (scores 15 or greater) as per the Short Arthritis Assessment Scale.
3. Significant cognitive deficits (scores <2) as per Ascertain Dementia 8 (AD8) questionnaire.
4. Significant visual field deficits as per the Humphrey Visual Field Analysis or significant uncorrected visual acuity deficits as per the Snellen Eye Chart.
5. Current treatment with anticoagulation medication
6. Parkinson's Disease or known Peripheral Neuropathy
7. Limitations to exercise related to cardiac, neurological or pulmonary diseases
8. Orthostatic hypotension
9. Severe osteoporosis defined by fracture history, BMD by DEXA (T score more than 2.5 standard deviations below controls in the last 2 years), or height loss of more than 3 cm
10. Current treatment with corticosteroids or aromatase inhibitor
11. Current treatment with seizure medication

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Test the efficacy of a wearable shoe sensor to detect initiation of abnormal gait patterns that increase the likelihood of falls | 1 hour; The entire protocol for testing the PD shoe is expected to be less than 2hours.
  Investigators will use pearson's correlation tests on gait variables (cadence, velocity, stride and step lengths) on Dynamic Gait Index that correlate with visual, proprioceptive and vestibular impairments and functional indicators of fall risk (e.g., Berg Balance Scale, Dynamic Gait Index, Activities Specific Balance Confidence questionnaire, Dizziness Handicap Inventory, Gaze Stabilization and Head Thrust Test) to determine variables that indicate an increased likelihood of falls.

SECONDARY OUTCOMES:
Assess effectiveness of a gait synchronized vibration system to the plantar surface in reducing fall risk. | 1 hour; The entire protocol for testing the PD shoe is expected to be less than 2hours.
  Investigators will measure the change in gait parameters (cadence, velocity, stride and step lengths) and performance on the Dynamic Gait Index with and without vibratory stimulus.

OTHER OUTCOMES:
ABC Confidence Scale | 30 Minutes
  Self administered 16 question assessment in which subjects are instructed to answer each question with a percentage of confidence that they will not fall while performing a given task from 0%-100%, with 0% being "not confident" and 100% being "confident". Scores 80% or higher indicate a high level of physical functioning, 50-80% indicate a moderate level of physical functioning and scores less than 50% indicate a low level of physical functioning. The cut off for participation in the study will be <80%
Ascertain Dementia 8 (AD8) | 15 Minutes
  Eight questions requiring the participant to indicate whether there has been a recent change in memory, problem-solving abilities, orientation and ability to perform daily activities with either "yes" or "no" answers. The numbers of "yes" answers are totaled to obtain the AD8 score. Scores of 0-1 are considered normal cognition, while scores greater than 2 are suggestive of cognitive impairment. The cut off for participation in the study will be < 2
Balance Master | 15 Minutes
  Subjects will ask to stand on the Balance Master system to gain objective information regarding integration of sensory and visual input and proprioception in a static or dynamic setting.
Berg Balance Scale (BBS) | 20 Minutes
  of 14 tasks used to determine the participant's ability to balance in different functional situations. Each item is scored 0-4 for a maximum of 56 points. Scores 0-20 represent very high fall risk, 21-40 moderate fall risk and scores 41-56 indicate low fall risk. Item description includes: sitting to standing, standing unsupported, sitting unsupported, standing to sitting, transfers, standing with eyes closed, standing with feet together, reaching forward with outstretched arm, retrieving object from floor, turning to look behind, turning 360 degrees, placing alternate foot on stool, standing with one foot in front, standing on one foot. The cut off for participation in the study will be > 20.
Dizziness Handicap Inventory | 15 Minutes
  Self reported questionnaire designed to identify functional, physical or emotional difficulties subjects experience as a result of dizziness or unsteadiness. Subjects will answer the 25 item form with "yes" (4 points), "sometimes" (2 points) and "no" (0 points) for a maximum of 100 points. Scores 16-34 indicate a mild handicap, 36-52 a moderate handicap and scores 54 or greater indicate severe handicap. The cut off for participation in the study will be scores <16.
Dynamic Gait Index | 30 Minutes
  This test will evaluate an individual's impairments in ambulating under different circumstances to assess for fall risk. Subjects will be asked to walk under normal circumstances on level ground, walking as quickly as they can, walking with horizontal head turns, vertical head turns, stop and pivot, step over obstacles, step around obstacles and walking up stairs. Subjects will be scored out of a possible 24 points for the 8 domains awarding 3 points for normal ambulatory patterns, 2 points for mild impairments in performing exercises, 1 point for moderate impairments and 0 points for severe impairment. Scores less than or equal to 19 are predictive of falls whereas scores 22 or greater indicate safe ambulators. The cut off for participation in the study will be scores <22
Gaze Stabilization via the Head Thrust Test | 10 Minutes
  The subject's head is suddenly and rapidly rotated through a small range (15-30 degrees) and then stopped. The patient's task is to maintain fixation on a visual target. This is repeated to both sides. Individuals with normal vestibular function will be able to maintain visual fixation. Individuals with bilateral vestibular loss will demonstrate corrective saccades following the head thrust test in both directions. Individuals with unilateral vestibular loss will demonstrate corrective saccades after head rotation towards the side of decreased function. The cut off for participation in the study will be any corrective saccades following cessation of head rotation.
Humphrey Visual Field Testing | 10 Minutes
  This test will be used to evaluate each subject's peripheral vision for visual field deficits. Subjects will be allowed to wear their normal corrective lenses if applicable. Individuals with significant visual field deficits will not be enrolled in the study.
Six Minute Walk Test | 18 Minutes
  Subjects will be asked to walk as far as they can over a period of six minutes as rapidly as they can. We will evaluate the difference between distances walked at baseline with regular foot wear, while wearing the shoe without vibratory stimulus to assess gait parameters using the shoe sensor and finally while wearing the shoe with vibratory stimulus turned on.
Short Arthritis Assessment Scale (SAS) | 1 Minute
  4 Question visual analog scale in which participants score from 0-10 how their arthritic pain impacts their life, for a total score of 40 points. The questionnaire asks participants to score how much pain they have experienced during the past week from 0 (no pain) to 10 (severe pain), followed by how much difficulty is experienced in physical functioning during stair navigation and shopping ranked from 0 (no difficulty) to 10 (extreme difficulty), then overall how well they are coping with their arthritis pain and how they feel they are doing from 0 (very well) to 10 (very poor). Scores below 7 show minimal arthritic pain and scores cutting at 15 and 25 show increasing severity of symptoms. The cut off for participation in the study will be <=7.
Snellen Eye Chart | 1 Minute
  Subjects will be screened for uncorrected visual acuity deficits using their normal corrective lenses if applicable. Individuals with uncorrected visual acuity less than 20/40 will not be enrolled in the study
Timed Up and Go Test | 2 Minutes
  Subjects, wearing regular footwear, will begin in a seated position in an arm chair and are instructed to rise, walk three meters and return to the chair and assume the seated position once more. The examiner will begin timing the patient on the word "go" and will stop time when the patient completes the exercise. A score greater than 15 seconds in this assessment indicates an increased risk for falls.
Video Documentation | 6 Minutes
  Subjects will be videotaped during their performance in the Six Minute Walk Test and the Dynamic gait index to visually assess and document any changes in gait parameters such as cadence, velocity, stride and step lengths under conditions of baseline level walking and with and without vibratory stimulus. The videotaping procedures will focus on the subject's lower extremities but may include their face in order to fully capture the gait

CONTACTS AND LOCATIONS:
Overall Officials: Preeti Raghavan, M.D., Principal Investigator — New York University Medical School

IPD SHARING:
Plan to Share IPD: No
Study has been withdrawn